CLINICAL TRIAL: NCT01088919
Title: A Phase 1, Open Label, Randomized, Crossover, Drug Interaction Study of the Pharmacokinetics of ASP1941 and Pioglitazone Hydrochloride After Separate and Concomitant Administration to Healthy Adult Subjects
Brief Title: A Study to Characterize the Effect on the Pharmacokinetics of ASP1941 and Pioglitazone Hydrochloride When Given Together to Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sr Manager Clinical Trials Registry, Astellas Pharma Global Development
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 1941-CL-0060
Record Dates: First submitted 2010-03-04; First posted 2010-03-18 (Estimated); Last update posted 2010-04-16 (Estimated); Status verified 2010-04

CONDITIONS: Healthy; Pharmacokinetics of ASP1941
Keywords: ASP1941; Actos; pioglitazone hydrochloride
MeSH Terms: interventions — ipragliflozin; Pioglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Dosing Regimen 1 (Experimental)
  Interventions: Drug: ASP1941; Drug: pioglitazone hydrochloride
- Dosing Regimen 2 (Experimental)
  Interventions: Drug: ASP1941; Drug: pioglitazone hydrochloride
- Dosing Regimen 3 (Experimental)
  Interventions: Drug: ASP1941; Drug: pioglitazone hydrochloride
- Dosing Regimen 4 (Experimental)
  Interventions: Drug: ASP1941; Drug: pioglitazone hydrochloride

INTERVENTIONS:
Drug: ASP1941 — oral tablet
Drug: pioglitazone hydrochloride — oral tablet
  Other Names: Actos

SUMMARY:
The purpose of this study is to evaluate pharmacokinetics, pharmacodynamics and safety following the administration of ASP1941 and pioglitazone hydrochloride in multiple and single doses.

DETAILED DESCRIPTION:
All subjects will be enrolled at one center and confined to the unit for up to 23 days. Subjects will be dosed in the fasting state in one of the four groups.

ELIGIBILITY:
Inclusion Criteria:

* The subject weighs at least 50 kg, and has a body mass index (BMI) of 18 to 32 kg/m2 inclusive
* The subject's 12-lead electrocardiogram (ECG) results are normal
* The female subject must be at least two years postmenopausal, surgically sterile or practicing effective birth control and not pregnant or lactating
* The male or female subject agrees to practice highly effective birth control from Screening until 7 days post last dose

Exclusion Criteria:

* The subject has a history or evidence of any clinically significant (as determined by the investigator) cardiovascular, endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, renal, and/or other major disease or malignancy (excluding non-melanoma skin cancer)
* The subject has any condition possibly affecting drug absorption (e.g., gastrectomy)
* The subject has history of consuming more than 14 units of alcoholic beverages per week within 6 months prior to screening or has a history of alcoholism or drug/chemical/substance abuse within past 2 years prior to screening or the subject tests positive for alcohol or drugs of abuse
* The subject has/had febrile illness or symptomatic, viral, bacterial (including upper respiratory infection), or fungal (non-cutaneous) infection within 1 week prior to clinic check in
* The subject has a supine mean systolic blood pressure < 90 or > 160 mmHg and a mean diastolic blood pressure < 50 or > 90 mmHg, or pulse rate higher than 100 beats per min (bpm)
* The subject has a 12-lead ECG demonstrating QTc >470 msec (female) or >450 msec (male)
* The subject is known positive for human immunodeficiency virus (HIV) antibody
* The subject has a positive test for tuberculosis (TB), hepatitis C antibody, or positive for hepatitis B antigen (HBsAg)
* The subject has used prescription or non-prescription drugs within 2 weeks or 5 half-lives (whichever is longer) or complementary and alternative medicines (CAM) within 14 days prior to study drug administration (excluding oral contraceptives, hormone replacement therapy [HRT], and acetaminophen)
* The subject has had any significant blood loss, donated one unit (450 mL) of blood or more, or received a transfusion of any blood or blood products within 60 days or donated plasma within 7 days prior to clinic admission

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2009-11; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic variables assessment through analysis of blood samples | Day 1 and up to Day 21

SECONDARY OUTCOMES:
Pharmacodynamic variables assessment through analysis of blood and urine samples | Day -1 and up to Day 17
Safety assessed by recording of adverse events, laboratory assessments, electrocardiograms (ECGs), vital signs and physical examinations | Day 1 through scheduled group check out (Day 13 and up to Day 21) or early termination

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Director — Astellas Pharma Global Development
Locations (1):
- Miami, Florida, United States